CLINICAL TRIAL: NCT01287494
Title: Collaborative Care for Depressed Elders in China
Brief Title: Depression Care Management for Depressed Elders in China Primary Care
Acronym: DCM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Zhejiang University, Zhejiang University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: DCM in China
Record Dates: First submitted 2011-01-27; First posted 2011-02-01 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Depression
Keywords: elderly; care management; primary care
MeSH Terms: conditions — Depression | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Depression Care Management (Experimental): DCM Intervention for Depressed Elders in Primary Care
  * Treatment guidelines (TG): Eight weeks treatment with Sertraline, another 8 weeks treatment augmentation with Bupropion if patients fail to respond in the initial trial, For more complicated cases, the transfer to psychiatrists is indicated.
  * Care managers: Screening, Adherence support, psychoeducation and communication.
  * Psychiatric Consultation
  Interventions: Drug: Sertraline
- Care as Usual (No Intervention)

INTERVENTIONS:
Drug: Sertraline — dosage form: Capsule dosage: 50-200mg/d frequency: once per day duration: 16 weeks
  Other Names: Zoloft
  Arms: Depression Care Management

SUMMARY:
Using a randomized controlled design, the investigators will examine whether the DCM is an effective treatment for patients with late life depression in urban China. Our specific aims are: (1) to determine whether the DCM intervention results in improved outcomes compared with CAU at both the provider (e.g., greater adherence to quality indicators) and patient levels (e.g., greater reduction in depressive symptoms); and (2) to compare DCM with CAU with regard to a range of outcomes in other pertinent domains, both at the provider (e.g., improvements in knowledge/attitudes) and patient (e.g., functioning, satisfaction) levels. The study will take place in 16 primary care clinics (PCCs) randomly assigned to deliver either DCM or CAU (8 clinics each) to 320 patients (aged≥60 years) with major depression (20/clinic; n=160 in each treatment condition). In the DCM arm, PCPs will prescribe 16 weeks of antidepressant medication according to the TG protocol. CMs monitor the progress of treatment and side effects, educate patients/family, and facilitate communication between providers; psychiatrists will provide weekly group psychiatric consultation and CM supervision. Patients in both DCM and CAU arms will be assessed by clinical research coordinators at baseline, 4, 8, 12, 18, and 24 months. HDRS, MMSE, CAS, SF-12, Treatment Stigma and the Client Satisfaction Questionnaire will be used to assess patients' outcomes; and clinic practices, attitudes/knowledge, and satisfaction will be providers' outcomes.

DETAILED DESCRIPTION:
* At the patient level: The investigator will gather information about age, gender, education, marital status, living conditions and satisfaction with their economic status, as well as systematic information on suicidal ideation,, psychopathology, medical health, cognitive function, quality of life and stigma and satisfaction for the treatment.
* At the provider level: the objective of research measures at the provider level is to gather social-demographic data such as age, gender, education, marital status, clinical experience among physicians in the participating PCCs as well as systematic information on their attitudes/knowledge regarding depression and clinical practices with the treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years old
* Community-dwelling residences
* Capable of independent communication
* Mini-Mental State Examination (MMSE) score ≥ 18

Exclusion Criteria:

* Incapable of giving written informed consent to this study
* Acute high suicide risk at baseline assessment
* Psychosis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2010-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
the DCM intervention results in improved outcomes compared with CAU at both the provider (e.g., greater adherence to quality indicators) and patient levels (e.g., greater reduction in depressive symptoms) | 16 weeks
  16 weeks treatment with Sertraline and following up 2 years

SECONDARY OUTCOMES:
compare DCM with CAU with regard to a range of outcomes in other pertinent domains, both at the provider (e.g., improvements in knowledge/attitudes) and patient (e.g., functioning, satisfaction) levels | 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Ju Zhang, PhD, Study Director — Zhejiang University
Locations (1):
- Zhejiang Univeristy, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Chen S, Chiu H, Xu B, Ma Y, Jin T, Wu M, Conwell Y. Reliability and validity of the PHQ-9 for screening late-life depression in Chinese primary care. Int J Geriatr Psychiatry. 2010 Nov;25(11):1127-33. doi: 10.1002/gps.2442. PMID 20029795
- [Derived] Chen S, Conwell Y, He J, Lu N, Wu J. Depression care management for adults older than 60 years in primary care clinics in urban China: a cluster-randomised trial. Lancet Psychiatry. 2015 Apr;2(4):332-9. doi: 10.1016/S2215-0366(15)00002-4. Epub 2015 Mar 31. PMID 26360086
- [Derived] Chen S, Conwell Y, Xu B, Chiu H, Tu X, Ma Y. Depression care management for late-life depression in China primary care: protocol for a randomized controlled trial. Trials. 2011 May 13;12:121. doi: 10.1186/1745-6215-12-121. PMID 21569445